CLINICAL TRIAL: NCT00761735
Title: Assessment of the Safety, Efficacy, Tolerability and Pharmacokinetics of PEG-Intron® Plus REBETOL® in Pediatric Patients With Chronic Hepatitis C
Brief Title: 5 Year Long-term Follow up in Pediatric Participants Who Received PegIntron Plus Rebetol in P02538 Part I (P02538 Pt 2)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P02538: Part 2; 2004-000558-22 (EudraCT Number)
Record Dates: First submitted 2008-09-05; First posted 2008-09-29 (Estimated); Results first posted 2013-12-17 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — peginterferon alfa-2b; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PEG-IFN + RBV: LTFU (Other): Pediatric participants who completed treatment with peginterferon alfa-2b (PEG-IFN) plus ribavirin (RBV) in P02538 Part 1 of this study (NCT00104052) were enrolled in a 5-year Long Term Follow-Up (LTFU) during P02538 Part 2 (NCT00761735). No study treatment was administered in Part 2.
  Interventions: Biological: Peginterferon alfa-2b; Drug: Ribavirin

INTERVENTIONS:
Biological: Peginterferon alfa-2b — In the previous treatment protocol (P02538 Part 1), peginterferon alfa-2b was administered at a dose of 60 μg/m^2 by subcutaneous injection weekly for up to 48 weeks. No treatment was administered on the current follow-up study (P02538 Part 2).
  Other Names: PEG-Intron®
Drug: Ribavirin — In the previous treatment protocol (P02538 Part 1), ribavirin was administered at a dose of 15 mg/kg/day orally in two divided doses for up to 48 weeks. No treatment was administered on the current follow-up study (P02538 Part 2).
  Other Names: REBETOL®

SUMMARY:
Study P02538 Part 2 is a 5-year long term follow-up (LTFU) study in pediatric participants who were treated with at least one dose of peginterferon alfa-2b (PEG-IFN) and ribavirin (RBV) and who completed the follow-up in the P02538 Part 1 study (NCT00104052). No study drug therapy will be administered during the P02538 Part 2 study. Durability of virologic response will be assessed for participants who attained sustained virologic response (SVR) in Part I of this study by performing annual Hepatitis C Virus ribonucleic acid (HCV-RNA) testing. In addition, this study will characterize long-term safety in all participants who received PEG-IFN plus RBV treatment.

DETAILED DESCRIPTION:
During the Part 2 LTFU, participants will be evaluated at Years 1, 2, 3, 4, and 5. Each participant's first LTFU visit will be scheduled approximately 1 year after the post-treatment Follow-up Week 24 visit in Part 1 of this study (NCT00104052).

ELIGIBILITY:
Inclusion Criteria:

* Informed consent must be obtained from the participant or the participant's parent or legal guardian prior to any long-term follow-up study-related procedures. According to local laws and/or IRB/IEC requirements, participants may also need to provide written assent.
* The participant must have received at least one dose of peginterferon alfa-2b and ribavirin in the Protocol No. P02538 study.
* The participant must have completed the 24-week post-treatment follow-up in the P02538 Part 1 study. All participants whether sustained responders, relapsers, or nonresponders are eligible to participate.

Exclusion Criteria:

* Concurrent participation in any other clinical study.
* Retreatment with any antiviral or immunomodulatory drug for chronic hepatitis C after completion of, or discontinuation from, the treatment phase of the P02538 Part 1 study.
* Any condition that in the opinion of the Investigator would make the participant unsuitable for enrollment.

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 94 (Actual)
Dates: Start 2007-07; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Wirth S, Ribes-Koninckx C, Calzado MA, Bortolotti F, Zancan L, Jara P, Shelton M, Kerkar N, Galoppo M, Pedreira A, Rodriguez-Baez N, Ciocca M, Lachaux A, Lacaille F, Lang T, Kullmer U, Huber WD, Gonzalez T, Pollack H, Alonso E, Broue P, Ramakrishna J, Neigut D, Valle-Segarra AD, Hunter B, Goodman Z, Xu CR, Zheng H, Noviello S, Sniukiene V, Brass C, Albrecht JK. High sustained virologic response rates in children with chronic hepatitis C receiving peginterferon alfa-2b plus ribavirin. J Hepatol. 2010 Apr;52(4):501-7. doi: 10.1016/j.jhep.2010.01.016. Epub 2010 Feb 4. PMID 20189674

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 107 participants who enrolled in Part 1 of this study and were potentially eligible for the Part 2 Long Term Follow-up (LTFU), 94 participants enrolled in the current LTFU study (Part 2).
Period: Overall Study
Arm/Group | PEG-IFN + RBV: LTFU
Started | 94
Completed | 80
Not Completed | 14
Not completed — Lost to Follow-up | 6
Not completed — Withdrawal by Subject | 6
Not completed — Non-compliance with protocol | 1
Not completed — Administrative | 1

BASELINE CHARACTERISTICS:
Arm/Group | PEG-IFN + RBV: LTFU
Number analyzed (Participants) | 94
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.9 (3.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49
  Male | 45

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Relapsed At End of LTFU Year 5
Description: Relapse was defined as Hepatitis C Virus ribonucleic acid (HCV-RNA) that was above the lower limit of quantitation at Year 5 of the LTFU.
Time Frame: Part 2 LTFU Year 5
Population: Of 94 participants entering the P02538 Part 2 LTFU, 63 participants had achieved sustained virologic response (SVR) while in Part 1 of the study. 54 of these 63 participants completed 5 years of LTFU and were evaluated for relapse.
Measure: Number; unit: participants
Groups:
- PEG-IFN + RBV: LTFU (All): Pediatric participants who completed treatment with peginterferon alfa-2b (PEG-IFN) plus ribavirin (RBV) in P02538 Part 1 of this study (NCT00104052) were enrolled in a 5-year Long Term Follow-Up (LTFU) during P02538 Part 2 (NCT00761735). No study treatment was administered in Part 2.
Arm/Group | PEG-IFN + RBV: LTFU (All)
Number analyzed (Participants) | 54
participants | 0

2. Primary Outcome: Mean Height Percentiles of Participants Over LTFU
Description: To determine long-term effects of the Part 1 treatment on height, changes in height during the Part 2 LTFU were evaluated using height percentiles based on 2000 Center For Disease Control growth charts for the general population.
Time Frame: Part 1 Pre-treatment Baseline, Part 2 LTFU Year 1, Part 2 LTFU Year 2, Part 2 LTFU Year 3, Part 2 LTFU Year 4, Part 2 LTFU Year 5, Last Available LTFU Visit (up to 5 years)
Population: All participants enrolled in the P02538 Part 2 LTFU were evaluated in this analysis.
Measure: Mean (Standard Deviation); unit: percentile
Groups:
- PEG-IFN + RBV: LTFU (24 Weeks): Pediatric participants who completed 24 weeks of treatment with PEG-IFN plus RBV in P02538 Part 1 of this study (NCT00104052) were enrolled in a 5-year LTFU during P02538 Part 2 (NCT00761735). No study treatment was administered in Part 2.
- PEG-IFN + RBV: LTFU (48 Weeks): Pediatric participants who completed 48 weeks of treatment with PEG-IFN plus RBV in P02538 Part 1 of this study (NCT00104052) were enrolled in a 5-year LTFU during P02538 Part 2 (NCT00761735). No study treatment was administered in Part 2.
Arm/Group | PEG-IFN + RBV: LTFU (24 Weeks) | PEG-IFN + RBV: LTFU (48 Weeks)
Number analyzed (Participants) | 46 | 48
percentile
  Part 1 Pre-treatment Baseline | 48.94 (27.38) | 52.5 (29.98)
  LTFU Year 1 (n=40, n=44) | 49.21 (29.03) | 43.37 (27.87)
  LTFU Year 2 (n=39, n=39) | 50.56 (29.18) | 46.24 (29.19)
  LTFU Year 3 (n=39, n=44) | 48.05 (28.38) | 46.00 (28.24)
  LTFU Year 4 (n=40, n=38) | 49.62 (30.87) | 45.27 (29.44)
  LTFU Year 5 (n=38, n=42) | 47.61 (29.57) | 43.51 (27.57)
  Last Available LTFU Visit (n=46, n=48) | 45.96 (30.45) | 43.56 (27.19)

3. Primary Outcome: Mean Weight Percentiles of Participants Over LTFU
Description: To determine long-term effects of the Part 1 treatment on weight, changes in weight during the Part 2 LTFU were evaluated using weight percentiles based on 2000 Center For Disease Control growth charts for the general population.
Time Frame: as for outcome 2
Population: All participants enrolled in the P02538 Part 2 LTFU were evaluated in this analysis.
Measure: Mean (Standard Deviation); unit: percentile
Arm/Group | PEG-IFN + RBV: LTFU (24 Weeks) | PEG-IFN + RBV: LTFU (48 Weeks)
Number analyzed (Participants) | 46 | 48
percentile
  Part 1 Pre-treatment Baseline | 52.5 (26.83) | 58.56 (30.56)
  LTFU Year 1 (n=40, n=44) | 53.62 (26.75) | 56.38 (30.55)
  LTFU Year 2 (n=39, n=39) | 51.73 (26.89) | 52.03 (30.47)
  LTFU Year 3 (n=39, n=44) | 53.18 (29.12) | 54.26 (30.37)
  LTFU Year 4 (n=40, n=38) | 51.75 (28.90) | 49.50 (30.37)
  LTFU Year 5 (n=38, n=42) | 51.16 (27.16) | 53.12 (31.38)
  Last Available LTFU Visit (n=46, n=48) | 50.15 (28.44) | 55.53 (30.67)

4. Primary Outcome: Mean Body Mass Index (BMI) Percentiles of Participants Over LTFU
Description: To determine long-term effects of the Part 1 treatment on BMI, changes in BMI during the Part 2 LTFU were evaluated using BMI percentiles based on 2000 Center For Disease Control growth charts for the general population.
Time Frame: as for outcome 2
Population: All participants enrolled in the P02538 Part 2 LTFU were evaluated in this analysis.
Measure: Mean (Standard Deviation); unit: percentile
Arm/Group | PEG-IFN + RBV: LTFU (24 Weeks) | PEG-IFN + RBV: LTFU (48 Weeks)
Number analyzed (Participants) | 46 | 48
percentile
  Part 1 Pre-treatment Baseline | 50.4 (29.63) | 59.76 (31.52)
  LTFU Year 1 (n=40, n=44) | 51.15 (30.27) | 59.91 (31.55)
  LTFU Year 2 (n=39, n=39) | 48.11 (29.59) | 52.89 (30.82)
  LTFU Year 3 (n=39, n=44) | 52.14 (31.00) | 54.96 (30.89)
  LTFU Year 4 (n=40, n=38) | 48.44 (30.46) | 48.69 (31.52)
  LTFU Year 5 (n=38, n=42) | 48.61 (29.72) | 52.34 (31.87)
  Last Available LTFU Visit (n=46, n=48) | 48.79 (29.40) | 55.38 (31.48)

5. Primary Outcome: Mean Age at Attained Tanner Stages (Sexual Maturity) at End of LTFU (Last Observation) By Gender
Description: The Tanner Stage (TS) defines physical measurements of sexual development based on external primary and secondary sex characteristics. Female participants are evaluated for breast development and pubic hair distribution and male participants are evaluated for genital development and pubic hair distribution, based on a 5-stage ordinal scale ranging from TS 1 (prepubertal/preadolescent characteristics) to TS 5 (mature or adult characteristics). Mean ages for attaining each TS in the normal population have been previously established based on measuring correlating reproductive hormone levels, and are expressed in years as follows for females (F) and males (M): TS 1= 7.1 (F+M); TS 2= 10.5 (F), 12.1 (M); TS 3= 11.6 (F), 13.6 (M); TS 4=, 12.3 (F), 15.1 (M); TS 5= 14.5 (F), 18 (M). To assess sexual maturation at the end of the LTFU (last observation), females and males were staged and the mean age at each TS attained was reported.
Time Frame: Last assessment of the Part 2 LTFU (up to 5 years)
Population: All participants enrolled in the P02538 Part 2 LTFU with non-missing Tanner Stage data at the last observation (up to Year 5 of the LTFU) were analyzed.
Measure: Mean (Standard Deviation); unit: years
Groups:
- PEG-IFN + RBV: LTFU (Female): Female pediatric participants who completed treatment with PEG-IFN plus RBV in P02538 Part 1 of this study (NCT00104052) were enrolled in a 5-year LTFU during P02538 Part 2 (NCT00761735). No study treatment was administered in Part 2.
- PEG-IFN + RBV: LTFU (Male): Male pediatric participants who completed treatment with PEG-IFN plus RBV in P02538 Part 1 of this study (NCT00104052) were enrolled in a 5-year LTFU during P02538 Part 2 (NCT00761735). No study treatment was administered in Part 2.
Arm/Group | PEG-IFN + RBV: LTFU (Female) | PEG-IFN + RBV: LTFU (Male)
Number analyzed (Participants) | 41 | 42
years
  Age of TS 1 participants (n=4, n=5) | 9.75 (1.13) | 11.00 (0.80)
  Age of TS 2 participants (n=5, n=3) | 11.86 (0.78) | 12.53 (1.27)
  Age of TS 3 participants (n=7, n=1) | 15.26 (4.64) | 13.60 (0)
  Age of TS 4 participants (n=4, n=6) | 16.00 (4.31) | 14.75 (1.47)
  Age of TS 5 participants (n=21, n=27) | 17.37 (2.71) | 19.18 (2.48)

ADVERSE EVENTS:
Time Frame: 5 years, starting after the Part 1 post-treatment Follow-up Week 24 visit
Description: Only serious adverse events were collected during this 5 year LTFU study.
Arm/Group | PEG-IFN + RBV: LTFU
Serious Adverse Events (participants affected / at risk) | 3/94
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PEG-IFN + RBV: LTFU (N=94)
Talipes (Congenital, familial and genetic disorders) | 1 (3)
Appendicitis (Infections and infestations) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor shall have editorial rights with respect to publications, abstracts, slides, and manuscripts and the right to review and comment on the data analysis and presentation with regard to (1) proprietary information that is protected, (2) the accuracy of the information contained in the publication, and (3) to ensure that the presentation is fairly balanced and in compliance with FDA regulations.